CLINICAL TRIAL: NCT05180396
Title: A Multicenter, Cross-sectional Study Evaluating the Symptoms, Clinical Follow-ups, Problems Encountered During the Course of the Disease, Disease Awareness and Treatment Compliance of Heart Failure Patients - AWARENESS HF-PD(Patient Diary)
Brief Title: A Study on Disease Awareness and Treatment Compliance of Heart Failure Patients
Acronym: AWARENESS-HF
Status: Completed | Type: Observational
Sponsor: AstraZeneca Turkey (Industry)
Collaborators: Klinar CRO (Other)
Responsible Party: Sponsor
Other Study IDs: K-J020
Record Dates: First submitted 2021-09-03; First posted 2022-01-06 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Questionnaire; ECHO; Prospective
MeSH Terms: conditions — Heart Failure | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases with the diagnosis of Heart Failure (Acute and Chronic): Application of a questionnaire consisting of different questions to patients.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Application of a study based questionnaire described in the protocol

SUMMARY:
The AWARENESS HF-PD is a cross-sectional, multicenter, survey-based study. Cases who were admitted to the outpatient clinic and hospitalized with the diagnosis of Heart Failure (Acute and Chronic) will be included in the study.

DETAILED DESCRIPTION:
Data entry personnel to be assigned at the centers throughout the study will apply a questionnaire consisting of different questions to patients referred to them by clinicians with the diagnosis of HF. In addition, clinical features of HF from the current file of the cases (NYHA, comorbid conditions, comorbid diseases, blood pressure, heart rate, latest biochemistry (BNP/NTproBNP if available), hematology test results, most recent ECG, most recent echocardiography , coronary angiography report, if any) will be recorded. No additional examination/procedure will be performed for the study, only the data of the examinations requested by the clinician in routine clinical practice will be entered. A total of 200 patients from 3 centers will be included in this study over a six-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 and over
2. Patients diagnosed with acute or chronic heart failure
3. Patients who agreed to participate in the study

Exclusion Criteria:

1. Patients who stated that they did not agree to participate in the study
2. Patients who were not diagnosed with Heart Failure or whose diagnosis was changed or not confirmed during the index application
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases with the diagnosis of Heart Failure (Acute and Chronic) who were admitted to the outpatient clinic and hospitalized will be included in the study. It is planned to include 200 patients from 3 centers in this study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Demographics | 6 months
  At the end of the six-month recruitment period, demographic, symptoms, clinical follow-up status, d will be performed on all included patients.
Disease Information | 6 months
  At the end of the six-month recruitment period disease information, treatment compliance, and awareness assessment will be performed on all included patients.

SECONDARY OUTCOMES:
HF Risk Factors (BMI, Diabetes, Hypertension, HLP, Tobbaco Use, CV Hereditary, Menapause, MI History and History of CMP in family) | 6 months
  BMI, Diabetes, Hypertension, HLP, Tobbaco Use, CV Hereditary, Menapause, MI History and History of CMP in family
HF Percutaneous Intervention / Operation History (CRT, ICD, CRT-DI, Pacemaker, PKG, CABG and Heart Valve Operations) | 6 months
  CRT, ICD, CRT-DI, Pacemaker, PKG, CABG and Heart Valve Operations
HF Comorbidities (CAD, AF, COPD, CRF, Anemia, Iron Defficiency, Hypo- Hypertiroidy, OSAS) | 6 months
  (CAD, AF, COPD, CRF, Anemia, Iron Defficiency, Hypo- Hypertiroidy, OSAS
HF Laboratory Results (Glucose, BUN, Creatinine, GFR, Sodium, Potassium, Nt-ProBNP, ALT, AST, ALP, HS-CRP, cTN, Hemoglobine, WBC, Ferritine, TSAD, LDL, tryglyceride, ST3, GGT, INR, ST4) | 6 months
  Glucose, BUN, Creatinine, GFR, Sodium, Potassium, Nt-ProBNP, ALT, AST, ALP, HS-CRP, cTN, Hemoglobine, WBC, Ferritine, TSAD, LDL, tryglyceride, ST3, GGT, INR, ST4)
HF ECHO Results (EF, LA, SID, Mitral Defficiency, SPAB, DID, Septum, SEG Muscle Weakness, Trial Defficiency) | 6 Months
  (EF, LA, SID, Mitral Defficiency, SPAB, DID, Septum, SEG Muscle Weakness, Trial Defficiency)

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Akdeniz University Medical Faculty, Antalya
  - Kahramanmaraş Sütçü İmam University Medical Faculty, Kahramanmaraş
  - Mersin University Medical Faculty, Mersin

IPD SHARING:
Plan to Share IPD: No